CLINICAL TRIAL: NCT04757766
Title: VAP-PRO-C6. Effectiveness and Tolerability of Venoactive Drugs in Combination Therapy and Their Effect on the Overall Treatment Outcomes in Patients With Chronic Venous Diseases of CEAP Classes C6 in Real Clinical Practice
Brief Title: VAP-PRO-C6. Effectiveness and Tolerability of Venoactive Drugs in Combination Therapy in Patients With CVD (CEAP C6)
Acronym: VAP-PRO-C6
Status: Completed | Type: Observational
Sponsor: Servier Russia (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-05682-066-RUS
Record Dates: First submitted 2021-02-12; First posted 2021-02-17 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Chronic Venous Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: in daily everyday routine practice — The treatment of patients with chronic venous disease of CEAP classes C6 will be consistent with routine clinical practice, local label for the medical use of drugs and the specific clinical situation.

SUMMARY:
The VAP-PRO-C6 is a Russian multicenter observational program to be implemented at the routine visits and assessments. The program will include patients with chronic venous disease of CEAP classes C6. This program is planned to be carried out in Russia in 2021-2022.

DETAILED DESCRIPTION:
Aim of the program is to describe effectiveness and tolerability of systemic pharmacotherapy as a part of combination therapy and its effect on the overall treatment outcomes in patients with venous ulcers (CEAP classes C6) treated in real clinical settings.

The planned number of patients is 350.

The inclusion period lasts for 6 months. The treatment will be consistent with routine clinical practice, local label for the medical use of drugs and the specific clinical situation. The following objective methods will be used to assess the changes in the skin condition:

* measurement of the area of reference ulcer (using LesionMeter*) before and after the treatment;
* changes in status localis.
* The presence and location of venous reflux and/or occlusion. The study does not implicate any intervention to routine management of patients with chronic venous disease (CVD). In particular, in this study the parameters that are usually evaluated during the examination of patients with classes C6 CVD (CEAP) will be recorded. Special attention will be paid to evaluating changes of the area of referent VU using objective methods (measuring ulcer area using LesionMeter, time to ulcer healing).

  * LesionMeter is a generally available tool for measuring the venous ulcer area.

ELIGIBILITY:
Inclusion Criteria:

* CVD documented by venous DUS
* Age over 18 years
* Written informed consent is provided
* No treatment with venoactive drugs within 4 weeks prior to inclusion in the study
* Presence of a primary /active venous ulcer (class C6/ CEAP) that meets criteria for the referent ulcer
* No surgical intervention or procedure (including sclerotherapy) for CVD is planned

Exclusion Criteria:

* Withdrawal of the informed consent
* Pregnancy or willingness to become pregnant within at least 2 months after the end of the study
* Indications for surgery (including sclerotherapy)
* Serious violation or non adherence to the prescribed therapy/ regimen
* Use of prohibited drugs that can cause edema of lower extremities (calcium channel blockers, hormonal agents, NSAIDs, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with venous ulcers (CEAP classes C6) treated in real clinical settings
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The first Phlebological Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Venous Ulcers (CEAP Classes C6) Treated in Daily Clinical Practice: The treatment of patients with chronic venous disease of CEAP classes C6 will be consistent with routine clinical practice, local label for the medical use of drugs and the specific clinical situation Particular attention was paid to determining the reference Venous ulcer (VU) area dynamics using the objective methods (measurement of ulcer area and ulcer healing time).
Period: Overall Study
Arm/Group | Patients With Venous Ulcers (CEAP Classes C6) Treated in Daily Clinical Practice
Started | 349
Completed | 349
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: patients with venous ulcers (CEAP classes C6) treated in daily clinical practice
  The reference VU must meet the following criteria:
  * area is no less than 5 cm² but no more than 30 cm²,
  * phase 2 or 3 of the wound healing process,
  * location on the medial aspect of lower third of leg.
Arm/Group | Patients With Venous Ulcers (CEAP Classes C6) Treated in Daily Clinical Practice
Number analyzed (Participants) | 349
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 170
  >=65 years | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.95 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 233
  Male | 116
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 349

OUTCOME MEASURES:

1. Primary Outcome: Eeffectiveness of Systemic Pharmacotherapy as a Part of Combination Therapy
Description: % of patients with complete healing of the reference venous ulcer after 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Venous Ulcers (CEAP Classes C6) Treated in Daily Clinical Practice
Number analyzed (Participants) | 349
Participants | 243

2. Primary Outcome: Eeffectiveness of Systemic Pharmacotherapy
Description: % of patients with reduction in the CVD clinical class by CEAP classification
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Venous Ulcers (CEAP Classes C6) Treated in Daily Clinical Practice
Number analyzed (Participants) | 349
Participants | 247

3. Secondary Outcome: Healing of the Reference Venous Ulcers #1
Description: % of patients with healed reference VU after 3 months of treatment
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Venous Ulcers (CEAP Classes C6) Treated in Daily Clinical Practice
Number analyzed (Participants) | 349
Participants | 47

4. Secondary Outcome: Healing of the Reference Venous Ulcers at Visit 3 vs Baseline
Description: change in the area of reference VU in cm² (measured with LesionMeter application)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: cm²
Arm/Group | Patients With Venous Ulcers (CEAP Classes C6) Treated in Daily Clinical Practice
Number analyzed (Participants) | 349
cm² | 8.02 (4.06)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Patients With Venous Ulcers (CEAP Classes C6) Treated in Daily Clinical Practice
All-Cause Mortality (participants affected / at risk) | 0/349
Serious Adverse Events (participants affected / at risk) | 0/349
Other Adverse Events (participants affected / at risk) | 1/349
OTHER ADVERSE EVENTS (reported when occurring in more than 0.29% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Venous Ulcers (CEAP Classes C6) Treated in Daily Clinical Practice (N=349)
exacerbation of chronic gastritis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT04757766/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT04757766/ICF_001.pdf